CLINICAL TRIAL: NCT02194803
Title: Observation of Treatment Patterns With Lucentis and Real Life Ophthalmic Monitoring, Including Optional OCT in Approved Indications
Brief Title: Observation of Treatment Patterns With Lucentis in Approved Indications
Acronym: OCEAN
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002ADE18
Record Dates: First submitted 2014-06-11; First posted 2014-07-18 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Neovascular AMD, Visual Impairment Due to DME, Visual Impairment Due to Macular Oedema Secondary to Branch or Central RVO, Visual Impairment Due to CNV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort with routine OCT monitoring
- Cohort without routine OCT monitoring

SUMMARY:
A multicentre, open-label, non-interventional study to observe treatment patterns in patients with wet age-related macular degeneration (wAMD), with visual impairment due to diabetic macular edema (DME), due to macular edema following retinal vein occlusion (RVO) or due to chorioidal neovascularization following pathologic myopia (mCNV) with repeated intravitreal injections of Lucentis® (Ranibizumab) including optional OCT monitoring over a 24 months observational period under real life conditions.

ELIGIBILITY:
Inclusion criteria:

* Presence of

  * neovascular (wet) age-related macular degeneration (AMD),
  * visual impairment due to diabetic macular oedema (DME),
  * visual impairment due to macular oedema secondary to retinal vein occlusion (branch RVO or central RVO) or
  * visual impairment due to choroidal neovascularisation (CNV) secondary to pathologic myopia (PM)
* Patients for whom a therapy with Lucentis® is medically indicated.
* Written patients informed consent.

Exclusion criteria:

* As described in the SmPC.
* Preceding intravitreal treatment of the study eye with anti-VEGF drugs in the last three months before enrollment
* Preceding intravitreal treatment of the study eye with steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients suffering from neovascular eye pathology in real life setting for whom a therapy with Lucentis® is recommended by the treating physician in line with approved indications. Warnings and contraindications have to be taken into account according to the summary of product characteristics (SmPC).
Sampling Method: Probability Sample
Enrollment: 5778 (Actual)
Dates: Start 2011-12-08 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Visual Acuity (VA) to Month 12 | Baseline, Month 12
  Visual Acuity is measured either with ETDRS Scores, Snellen or decimal Scale according to routine clinical practice. Measurements are transferred to LogMAR for statistical analysis. LogMAR is defined as logarithm of the minimum angle of resolution.
Change from Baseline in Visual Acuity (VA) to Month 24 | Baseline, Month 24
  Visual Acuity is measured either with ETDRS Scores, Snellen or decimal Scale according to routine clinical practice. Measurements are transferred to LogMAR for statistical analysis. LogMAR is defined as logarithm of the minimum angle of resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Tübingen, Germany

REFERENCES:
- [Derived] Spital G, Schmitz-Valckenberg S, Muller B, Liczenczias E, Chang P, Heimes-Bussmann B, Ziemssen F, Liakopoulos S; ORCA study group. Interpretation of SD-OCT imaging data in real-life conditions versus standardized reading centre analysis in eyes with diabetic macular oedema or macular oedema secondary to retinal vein occlusion: 24-month follow-up of the ORCA study. Graefes Arch Clin Exp Ophthalmol. 2025 Jan;263(1):131-139. doi: 10.1007/s00417-024-06579-7. Epub 2024 Sep 19. PMID 39294392
- [Derived] Liakopoulos S, Spital G, Brinkmann CK, Schick T, Ziemssen F, Voegeler J, Koch M, Kirchhof B, Holz FG, Pauleikhoff D, Schmitz-Valckenberg S. ORCA study: real-world versus reading centre assessment of disease activity of neovascular age-related macular degeneration (nAMD). Br J Ophthalmol. 2020 Nov;104(11):1573-1578. doi: 10.1136/bjophthalmol-2019-315717. Epub 2020 Feb 17. PMID 32066561
- [Derived] Ziemssen F, Wachtlin J, Kuehlewein L, Gamulescu MA, Bertelmann T, Feucht N, Voegeler J, Koch M, Liakopoulos S, Schmitz-Valckenberg S, Spital G; OCEAN study group. Intravitreal Ranibizumab Therapy for Diabetic Macular Edema in Routine Practice: Two-Year Real-Life Data from a Non-interventional, Multicenter Study in Germany. Diabetes Ther. 2018 Dec;9(6):2271-2289. doi: 10.1007/s13300-018-0513-2. Epub 2018 Oct 4. PMID 30288700
- [Derived] Ziemssen F, Feltgen N, Holz FG, Guthoff R, Ringwald A, Bertelmann T, Wiedon A, Korb C; OCEAN study group. Demographics of patients receiving Intravitreal anti-VEGF treatment in real-world practice: healthcare research data versus randomized controlled trials. BMC Ophthalmol. 2017 Jan 19;17(1):7. doi: 10.1186/s12886-017-0401-y. PMID 28103831
- [Derived] Ziemssen F, Bertelmann T, Hufenbach U, Scheffler M, Liakopoulos S, Schmitz-Valckenberg S. [Delayed treatment initiation of more than 2 weeks. Relevance for possible gain of visual acuity after anti-VEGF therapy under real life conditions (interim analysis of the prospective OCEAN study)]. Ophthalmologe. 2016 Feb;113(2):143-51. doi: 10.1007/s00347-015-0099-2. German. PMID 26201460